CLINICAL TRIAL: NCT02959736
Title: Validating the Music Therapy Assessment Tool for Awareness in Disorders of Consciousness (MATADOC) Against the Best Practice External Reference Standard
Brief Title: Validating the MATADOC Against Best Practice Standard External Reference Standard
Acronym: MATADOC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Temple University (Other)
Collaborators: National Rehabilitation Hospital, Dublin, Ireland (NRH) (Unknown); Royal Hospital for Neuro-disability (Other); Corewell Health West (Other)
Responsible Party: Sponsor
Other Study IDs: 23925
Record Dates: First submitted 2016-11-07; First posted 2016-11-09 (Estimated); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Brain Injuries
Keywords: Vegetative State (VS); Minimally Conscious State (MCS); Brain Injuries
MeSH Terms: conditions — Brain Injuries; Persistent Vegetative State | interventions — Music Therapy; Reoperation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- National Rehabilitation Hospital Dublin: Music Therapy (MATADOC)
  Interventions: Behavioral: MATADOC and CRS-R
- Spectrum: Music Therapy (MATADOC)
  Interventions: Behavioral: MATADOC and CRS-R
- Royal Hospital for Neuro-disability London: Music Therapy (MATADOC)
  Interventions: Behavioral: MATADOC and CRS-R

INTERVENTIONS:
Behavioral: MATADOC and CRS-R — Behavioural assessments for Disorders of Consciousness
  Other Names: Music Therapy and Coma Recovery Scale (Revised) or CRS-R

SUMMARY:
The purpose of this project is to further develop a standardized music-based measure used in music therapy with adults who have emerged from coma following profound brain injury, but are not able to demonstrate responsiveness to their environment due to complex clinical needs. Building on previous work, the project aims to strengthen the psychometric properties (e.g. concurrent validity, responsiveness) of the measure for its use with adults with profound brain damage.

DETAILED DESCRIPTION:
Adult patients with prolonged disorders of consciousness (PDOC), but who have not been diagnosed as Minimally Conscious or Vegetative State, will be recruited. All participants will be assessed using the Music Therapy Assessment Tool for Awareness in Disorders of Consciousness (MATADOC) standardized protocol. Assessment intervention will take place in four individual clinical contacts, over a 16 day period. Data will be collected using the MATADOC rating form and scored according to the MATADOC manual. Participants will concurrently be assessed with Coma Recovery Scale-Revised (CRS-R).

The MATADOC is implemented by Music Therapists who have been trained in its use and who are experienced in working with adults with PDOC. CRS-R data will be collected by members of the treatment team who are experienced or trained in its use. MATADOC and CRS-R assessors will remain blinded to the data collected.

Analysis will compare diagnostic outcomes of the two measures as well as explore the function of comparable items of each measure across similar domains (e.g. auditory, visual).

ELIGIBILITY:
Inclusion Criteria:

* Medically stable patients (i.e. not currently suspected of or under investigation for infection)who have a prolonged disorder of consciousness i.e. has persisted for longer than 4 weeks
* Between the ages of 18 and 70 years of age
* A diagnosis of awareness (i.e., VS, MCS or emergent) is not confirmed or is under investigation
* Fluent in English language comprehension as reported by the family

Exclusion Criteria:

* Known pre-morbid hearing impairments
* The patient has a previous diagnosis of musicogenic epilepsy
* The patient had previously refused music therapy intervention
* Patients with a suspected diagnosis of locked-in syndrome
* Non-fluent in English comprehension as reported by family.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults who have acquired profound brain damage resulting in prolonged disorders of consciousness (PDOC).
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Music Therapy Assessment Tool for Awareness in Disorders of Consciousness (MATADOC) | 16 days
  Music based protocol

SECONDARY OUTCOMES:
Coma Recovery Scale - Revised (CRS-R) | 16 days
  Behavioural rating scale

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Magee, PhD, Principal Investigator — Professor
Locations (1):
- Temple University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No